CLINICAL TRIAL: NCT05520970
Title: A Phase IIb, Multicenter, Observer-Blinded, Randomized, Placebo-Controlled Trial to Evaluate the Immunogenicity and Safety of the AdCLD-CoV19-1 in Healthy Adults Aged 19 Years Old and Above
Brief Title: Safety and Immunogenicity of COVID-19 Vaccine, AdCLD-CoV19-1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study early terminated based on the sponsor(manufacture)'s decision
Sponsor: Cellid Co., Ltd. (Industry)
Collaborators: International Vaccine Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IVI-AdCLD-CoV19-1
Record Dates: First submitted 2022-06-20; First posted 2022-08-30 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: COVID-19; Vaccines
MeSH Terms: conditions — COVID-19 | interventions — AdCLD-CoV19-1 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study is designed as observer-blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 2 doses of AdCLD-CoV19-1 (Experimental): Group 1 will receive 2 doses of AdCLD-CoV19-1
  Interventions: Biological: AdCLD-CoV19-1
- 1 dose of AdCLD-CoV19-1 (Experimental): Group 2 will receive 1 doses of AdCLD-CoV19-1 followed by 1 dose of placebo
  Interventions: Biological: AdCLD-CoV19-1
- Placebo (Placebo Comparator): Group 2 will receive 1 doses of placebo followed by 1 dose of AdCLD-CoV19-1 after an interim analysis
  Interventions: Biological: AdCLD-CoV19-1

INTERVENTIONS:
Biological: AdCLD-CoV19-1 — All 200 participants will receive 2 doses of investigational product by 2 months interval via intramuscular injection in the deltoid region

SUMMARY:
The immunogenicity and safety profiles of AdCLD-CoV19-1 (5.0×10^10 VP/dose) will be assessed for 1-dose or 2-dose regimen in SARS-CoV-2 seronegative healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy individual aged 19 years and above at consent.
2. Individual willing to provide written informed consent to participate study voluntarily.
3. Individuals who can be followed up during the study period and can comply with the study requirements.
4. Individual who agrees not to donate blood during the study participation
5. Females of childbearing potential with negative serum or urinary pregnancy test on the day of screening.
6. Females of childbearing potential who are using an effective birth control method for at least 4 weeks before the screening and during the study participation.

Exclusion Criteria:

1. Prior SARS-CoV-2 infection confirmed by a rapid antibody kit at screening.
2. History of receiving any vaccine (licensed or investigational) for SARS-CoV-2.
3. History of SARS-CoV-1 or MERS vaccination and treatment.
4. Individual determined to be clinically significantly abnormal by the screening outcome based on medical history, physical examination, laboratory evaluations (positive serological tests for Hepatitis B surface antigen (HBsAg), Hepatitis C antibody, and Human Immunodeficiency Virus (HIV) antibody), electrocardiogram (ECG) and Chest X-ray, and the clinical judgment of the investigator.
5. Individual who has received other vaccines from 4 weeks prior to the first dose of test vaccination or planned to receive any vaccine within 4 weeks of the last dose of the study vaccine.
6. Febrile illness (tympanic temperature ≥ 38°C) or acute illness with any clinically significant, respiratory symptoms (e.g., sore throat, cough, sputum) within 3 days prior to the study vaccination.
7. Known history or allergy to study vaccine components and/or excipients or other medications, or any other allergies deemed by the investigator to increase the risk of an adverse event if they were to participate in the trial (e.g., Guillain-Barre Syndrome).
8. Individual with major congenital abnormalities, which in the opinion of investigator may affect the participant's participation in the study.
9. Chronic use of systemic steroids (>10 mg/day prednisone equivalent for periods exceeding 14 days), cytotoxic or other immunosuppressive drugs within the past 6 weeks.
10. Any abnormality or chronic disease which in the opinion of the investigator might be detrimental to the safety of the participant and interfere with the assessment of the study objectives.

    ① Respiratory diseases: Asthma, Chronic Obstructive Lung Disease (COPD), active or latent tuberculosis which require medication, etc.

    ② Serious cardiovascular diseases: Congestive heart failure, coronary artery disease, myocardial infarction, uncontrolled hypertension, myocarditis, pericarditis, etc.

    ③ Neurologic diseases: Epilepsy, seizure within 3 years, migraine, stroke, encephalopathy, Guillain-Barre Syndrome, encephalomyelitis, acute transverse myelitis, etc.

    ④ Malignant cancer diagnosed within the past 5 years (skin basal cell and squamous cell carcinoma are excluded).

    ⑤ Immune function disorders, including auto-immune diseases and immunodeficiency diseases (known HIV infection or other immune function disorders)

    ⑥ Other hepatobiliary, renal, endocrine, urinary tract, muscular skeletal diseases which the investigator considers clinically significant
11. Individual with hereditary or idiopathic angioneurotic edema
12. Individuals with behavioral or cognitive impairment or psychiatric disease or neural disorders that, in the opinion of the investigator, could interfere with the participant's ability to participate in the trial.
13. Individual with splenectomy and transplantation (including solid organ and bone marrow).
14. Individual with past history of thrombocytopenia and/or thrombosis, myocarditis or pericarditis or any other significant cardiac condition.
15. Individual with a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time resulting in contraindication for IM injections/blood extractions (Those who receive low dose aspirin (less than 100mg/day) are not excluded).
16. Receipt of immunoglobulin or blood-derived products in the past 12 weeks or plan to receive during the study period.
17. Body mass index (BMI) ≥ 30 kg/m2.
18. As per Investigator's medical judgement, an individual could be excluded from the study in spite of meeting all inclusion/exclusion criteria mentioned above.
19. Any female participant who is lactating*, pregnant or planning for pregnancy** during the course of study period.
20. Individual concomitantly enrolled or scheduled to be enrolled in another trial.
21. Individual who is research staff involved with the clinical study or family/household members of research staff.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-08-19 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
Proportion of immediate adverse events (AE) | Within 30 minutes post each dose injection
  • Proportion of immediate AE within 30 minutes post each dose injection
Proportion of solicited local and systemic AE | Within 7 days (Days 0 - 6) post each dose injection
  • Proportion of solicited local and systemic AEs within 7 days post each dose injection. Local AEs at the site of injection: Pain, tenderness, erythema/redness, swelling, induration, pruritis. Systemic AEs: Fever, fatigue/general weakness, chill, headache, myalgia, arthralgia, diarrhea, nausea/vomiting, abdominal pain, mucocutaneous reaction/rash, urticaria, dizziness, cough, dyspnea.
Proportion of unsolicited AE | Within 28 days post each dose injection
  • Proportion of unsolicited AEs within 28 days post each dose injection. Unsolicited AEs are all other adverse events (those that do not fall under the categories of solicited AEs).
Proportion of SAE | Throughout the study end, an average of 14 months (12 months post second dose injection)
  • Proportion of any SAE from the vaccination throughout the entire study. An AE or suspected adverse reaction is considered "serious" if at any dose (including overdose): Results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is an important medical event that may jeopardize the participant or may require intervention to prevent one of the other outcomes listed above.
Proportion of Adverse Event Of Special Interest (AESI) | Throughout the study duration, an average of 14 months (12 months post second dose injection)
  • Proportion of any AESI from the vaccination throughout the entire study. AESI are categorized into 1) AESIs included because they are seen with COVID-19 Disease, 2) AESI included because they have a proven or theoretical association with immunization in general, 3) AESI included because they have a proven or theoretical association with specific vaccine platform(s).
Proportion of Medically-Attended Adverse Events (MAAE) | Throughout the study duration, an average of 14 months (12 months post second dose injection)
  • Proportion of any MAAE from the vaccination throughout the entire study. Medically-attended AEs are AEs with medically-attended visits including hospital, emergency room, or other visits to or from medical personnel for any reason. Routine study visits will not be considered medically attended visits.
Proportion of clinically significant changes in clinical safety laboratory parameters | At 1, 2 and 4 weeks post each dose injection
  Proportion of clinically significant changes in clinical safety laboratory parameters at 1, 2 and 4 weeks post each dose injection
Geometric Mean Titer of 1 and 2 doses of AdCLD-CoV19-1 from baseline to 2 weeks post second dose injection (Neutralizing antibody) | At 2 weeks post second dose injection
  Geometric Mean Titer (GMT) of neutralizing antibody to the SARS-CoV-2 measured by wild-type virus neutralization assay from baseline to 2 weeks post second dose injection, induced by 2 doses of AdCLD-CoV19-1 at 2-month interval and by 1 dose of AdCLD-CoV19-1 followed by 1 dose of placebo at 2-month interval
Geometric Mean Fold Rise of 1 and 2 doses of AdCLD-CoV19-1 from baseline to 2 weeks post second dose injection (Neutralizing antibody) | At 2 weeks post second dose injection
  Geometric Mean Fold Rise (GMFR) of neutralizing antibody to the SARS-CoV-2 measured by wild-type virus neutralization assay from baseline to 2 weeks post second dose injection, induced by 2 doses of AdCLD-CoV19-1 at 2-month interval and by 1 dose of AdCLD-CoV19-1 followed by 1 dose of placebo at 2-month interval
Proportion of participants achieving seroresponse of 1 and 2 doses of AdCLD-CoV19-1 from baseline to 2 weeks post second dose injection (Neutralizing antibody) | At 2 weeks post second dose injection
  Proportion of participants achieving seroresponse (SR defined as at least 4-fold increase from baseline) of wild-type virus neutralizing antibody titer from baseline to 2 weeks post second dose injection, induced by 2 doses of AdCLD-CoV19-1 at 2-month interval and by 1 dose of AdCLD-CoV19-1 followed by 1 dose of placebo at 2-month interval
GMT of 1 and 2 doses of AdCLD-CoV19-1 from baseline to 2 weeks post second dose injection (ELISA) | At 2 weeks post second dose injection
  GMT of SARS-CoV-2 Spike-binding ELISA IgG antibody from baseline to 2 weeks post second dose injection, induced by 2 doses of AdCLD-CoV19-1 at 2-month interval and by 1 dose of AdCLD-CoV19-1 followed by 1 dose of placebo at 2-month interval
GMFR of 1 and 2 doses of AdCLD-CoV19-1 from baseline to 2 weeks post second dose injection (ELISA) | At 2 weeks post second dose injection
  GMFR of SARS-CoV-2 Spike-binding ELISA IgG antibody from baseline to 2 weeks post second dose injection, induced by 2 doses of AdCLD-CoV19-1 at 2-month interval and by 1 dose of AdCLD-CoV19-1 followed by 1 dose of placebo at 2-month interval
Proportion of participants achieving seroresponse of 1 and 2 doses of AdCLD-CoV19-1 from baseline to 2 weeks post second dose injection (ELISA) | At 2 weeks post second dose injection
  Proportion of participants achieving seroresponse (SR defined as at least 4-fold increase from baseline) of SARS-CoV-2 Spike-binding ELISA IgG antibody from baseline to 2 weeks post second dose injection, induced by 2 doses of AdCLD-CoV19-1 at 2-month interval and by 1 dose of AdCLD-CoV19-1 followed by 1 dose of placebo at 2-month interval

SECONDARY OUTCOMES:
GMT of 1 and 2 doses of AdCLD-CoV19-1 from baseline to 1, 3, 6 months post first dose injection and at 1, 3, 6 and 12 months post second dose injection (Neutralizing antibody) | At 1, 3, 6 months post first dose injection and at 1, 3, 6 and 12 months post second dose injection
  GMT of neutralizing antibody to the SARS-CoV-2 measured by wild-type virus neutralization assay from baseline to and 1, 3, and 6 months post first dose injection, and at 1, 3, 6 and 12 months post second dose injection, induced by 1 and 2 doses of AdCLD-CoV19-1 respectively
GMFR of 1 and 2 doses of AdCLD-CoV19-1 from baseline to 1, 3, 6 months post first dose injection and at 1, 3, 6 and 12 months post second dose injection (Neutralizing antibody) | At 1, 3, 6 months post first dose injection and at 1, 3, 6 and 12 months post second dose injection
  GMFR of neutralizing antibody to the SARS-CoV-2 measured by wild-type virus neutralization assay from baseline to and 1, 3, and 6 months post first dose injection, and at 1, 3, 6 and 12 months post second dose injection, induced by 1 and 2 doses of AdCLD-CoV19-1 respectively
Proportion of participants achieving seroresponse of 1 and 2 doses of AdCLD-CoV19-1 from baseline to 1, 3, 6 months post first dose injection and at 1, 3, 6 and 12 months post second dose injection (Neutralizing antibody) | At 1, 3, 6 months post first dose injection and at 1, 3, 6 and 12 months post second dose injection
  Proportion of participants achieving seroresponse (SR defined as at least 4-fold increase from baseline) of wild-type virus neutralizing antibody titer from baseline to and 1, 3, and 6 months post first dose injection, and at 1, 3, 6 and 12 months post second dose injection, induced by 1 and 2 doses of AdCLD-CoV19-1 respectively
GMT of 1 and 2 doses of AdCLD-CoV19-1 from baseline to 1, 3, 6 months post first dose injection and at 1, 3, 6 and 12 months post second dose injection (ELISA) | At 1, 3, 6 months post first dose injection and at 1, 3, 6 and 12 months post second dose injection
  GMT of SARS-CoV-2 Spike-binding ELISA IgG antibody from baseline to 2 weeks, and 1, 3, and 6 months post first dose injection, and at 1, 3, 6 and 12 months post second dose injection induced by 1 and 2 doses of AdCLD-CoV19-1, respectively
GMFR of 1 and 2 doses of AdCLD-CoV19-1 from baseline to 1, 3, 6 months post first dose injection and at 1, 3, 6 and 12 months post second dose injection (ELISA) | At 1, 3, 6 months post first dose injection and at 1, 3, 6 and 12 months post second dose injection
  GMFR of SARS-CoV-2 Spike-binding ELISA IgG antibody from baseline to 2 weeks, and 1, 3, and 6 months post first dose injection, and at 1, 3, 6 and 12 months post second dose injection induced by 1 and 2 doses of AdCLD-CoV19-1, respectively
Proportion of participants achieving seroresponse of 1 and 2 doses of AdCLD-CoV19-1 from baseline to 1, 3, 6 months post first dose injection and at 1, 3, 6 and 12 months post second dose injection (ELISA) | At 1, 3, 6 months post first dose injection and at 1, 3, 6 and 12 months post second dose injection
  Proportion of participants achieving seroresponse (SR defined as at least 4-fold increase from baseline) of SARS-CoV-2 Spike-binding ELISA IgG antibody from baseline to 2 weeks, and 1, 3, and 6 months post first dose injection, and at 1, 3, 6 and 12 months post second dose injection induced by 1 and 2 doses of AdCLD-CoV19-1, respectively
Cell Mediated Immunity (CMI) of 1 and 2 doses of AdCLD-CoV19-1 from baseline to 2 weeks, 6 months post first dose injection and 2 weeks, 6 and 12 months post second dose injection (Proportion of responders by Interferon-γ (IFN-γ) ELISpot) | At 2 weeks, 6 months post first dose injection and 2 weeks, 6 and 12 months post second dose injection
  Proportion of responders as measured by Interferon-γ (IFN-γ) ELISpot from baseline to 2 weeks, 6 months post first dose injection and 2 weeks, 6 and 12 months post second dose injection induced by 1 and 2 doses of AdCLD-CoV19-1, respectively
Cell Mediated Immunity (CMI) of 1 and 2 doses of AdCLD-CoV19-1 from baseline to 2 weeks, 6 months post first dose injection and 2 weeks, 6 and 12 months post second dose injection (Median spot forming units by Interferon-γ (IFN-γ) ELISpot) | At 2 weeks, 6 months post first dose injection and 2 weeks, 6 and 12 months post second dose injection
  Median spot forming units as measured by Interferon-γ (IFN-γ) ELISpot from baseline to 2 weeks, 6 months post first dose injection and 2 weeks, 6 and 12 months post second dose injection induced by 1 and 2 doses of AdCLD-CoV19-1, respectively

OTHER OUTCOMES:
Number of virologically-confirmed COVID-19 cases and clinical features in AdCLD-CoV19-1 recipients during the study period | Throughout the study duration, an average of 14 months
  * Occurrences of confirmed COVID-19
  * Occurrence of symptomatic COVID-19
  * Occurrences of hospitalized COVID-19
  * Occurrence of severe COVID-19
  * Death associated with COVID-19
  * Severity of symptoms associated with symptomatic COVID-19 episode
GMT against the circulating strains, including the variants of concern from baseline to 2 weeks post second dose injection induced by AdCLD-CoV19-1 (Neutralizing antibody) | At 2 weeks post second dose injection
  GMT of neutralizing antibody to the circulating strains measured by wild-type virus neutralization assay from baseline to 2 weeks post second dose injection induced by AdCLD-CoV19-1
GMFR against the circulating strains, including the variants of concern from baseline to 2 weeks post second dose injection induced by AdCLD-CoV19-1 (Neutralizing antibody) | At 2 weeks post second dose injection
  GMFR of neutralizing antibody to the circulating strains measured by wild-type virus neutralization assay from baseline to 2 weeks post second dose injection induced by AdCLD-CoV19-1
Proportion of participants achieving seroresponse against the circulating strains, including the variants of concern from baseline to 2 weeks post second dose injection induced by AdCLD-CoV19-1 (Neutralizing antibody) | At 2 weeks post second dose injection
  Proportion of participants achieving seroresponse (SR defined as at least 4-fold increase from baseline) of wild-type virus neutralizing antibody titer from baseline to 2 weeks post second dose injection induced by AdCLD-CoV19-1

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - Korea University Ansan Hospital, Ansan
  - Catholic University Seoul St.Mary's Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Korea University Guro Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No